CLINICAL TRIAL: NCT05332015
Title: The Effect of Oral Hypotonic Hydration in Pregnant Women With Isolated Oligohydramnios: a Randomized Controlled Study
Brief Title: The Effect of Oral Hypotonic Hydration in Isolated Oligohydramnios
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Karadag, MD, Associate Professor, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4/2
Record Dates: First submitted 2022-03-31; First posted 2022-04-18 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Oligohydramnios
Keywords: Oligohydramnios; Hydrotherapy; Hypotonic hydrotherapy
MeSH Terms: conditions — Oligohydramnios | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral hydration with normal water (Active Comparator): Oral hydration with drinkable normal water daily additional 2 liters for 5 days
  Interventions: Other: Hypotonic (distilled) water
- Oral hydration with distilled water (Active Comparator): Oral hydration with distilled water daily 2 liters for 5 days
  Interventions: Other: Normal water

INTERVENTIONS:
Other: Hypotonic (distilled) water — orally given daily two liters of distilled water
  Arms: Oral hydration with normal water
Other: Normal water — orally given daily two liters of normal water
  Arms: Oral hydration with distilled water

SUMMARY:
OBJECTIVE: The primary objective of our study is to compare the effects of routine hydration with additional 2 liters of normal water versus orally 2 liters of distilled water on the amount of amniotic fluid.

HYPOTHESIS: İsolated oligohydramnios, secondary to depleted maternal intravascular volume, can be reversed better with orally hypotonic water.

DETAILED DESCRIPTION:
BACKGROUND: Olygohydramniosis is a condition in which amniotic fluid levels are lower than expected for gestational age. It is typically diagnosed by ultrasound examination and may be described qualitatively (e.g., reduced amniotic fluid volume) or quantitatively (e.g., amniotic fluid index ≤5 cm, single deepest pocket <2 cm). Water hydration aims to decrease maternal osmolality and sodium concentration, increase water flow osmotically from maternal blood to fetal amniotic fluid, and improve uteroplacental perfusion.

A meta-analysis comparing maternal hydration's effect reported that maternal intravenous hydration had good results on AFI in pregnancies with isolated oligohydramnios and hypotonic solutions were more effective than isotonic fluids(1). Maternal oral hydration may slightly increase amniotic fluid and is safer than intravenous fluid administration or amnioinfusion.

Reducing the osmolality in maternal blood with oral hypotonic and isotonic fluids helps to direct the placental water passage towards the fetus, to improve uteroplacental perfusion, and as a result, to increase the amount of amniotic fluid in pregnant women with isolated oligohydramnios. Osmolality is further reduced by maternal oral hypotonic fluid, thus improving the amount of amniotic fluid.

The study protocol was approved by the Local Ethics Committee, and written informed consent will be taken from patients entering the study. The sample size was calculated based on the "Maternal hydration increases amniotic fluid index" study of Kilpatrick et al.(2). When 1.5 cm increase in AFI is considered significant, with 90% power and type 2 error (alpha): 0.05, the sample size is 20 for each group, and it is planned to include 40 pregnant women in total.

I

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age (GA) 28-39 weeks (based on the last menstrual period and confirmed by the results of ultrasound or determined through early pregnancy sonography)
* Isolated oligohydramnios cases
* Amniotic fluid index ≤ 5
* No pregnancy complications such as preeclampsia, gestational hypertension
* Intact fetal membranes.

Exclusion Criteria:

* Presence of fetal complications (membrane rupture, presence of fetal anomaly, intrauterine growth restriction)
* Presence of maternal systemic disease (nephropathy, cardiac disease)
* Multiple pregnancies
* Conditions in which the amount of amniotic fluid cannot be accurately assessed (morbid obesity)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-08-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Reversal of Oligohydramnios Using AFV Measures | admission, day 7
  The change between the basal amniotic fluid index and the value on day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya Training and Research Hospital, Antalya, Muratpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gizzo S, Noventa M, Vitagliano A, Dall'Asta A, D'Antona D, Aldrich CJ, Quaranta M, Frusca T, Patrelli TS. An Update on Maternal Hydration Strategies for Amniotic Fluid Improvement in Isolated Oligohydramnios and Normohydramnios: Evidence from a Systematic Review of Literature and Meta-Analysis. PLoS One. 2015 Dec 11;10(12):e0144334. doi: 10.1371/journal.pone.0144334. eCollection 2015. PMID 26658482
- [Background] Kilpatrick SJ, Safford KL, Pomeroy T, Hoedt L, Scheerer L, Laros RK. Maternal hydration increases amniotic fluid index. Obstet Gynecol. 1991 Dec;78(6):1098-102. PMID 1945215